CLINICAL TRIAL: NCT04745286
Title: Effects of Small-dose S-ketamine on Anesthesia-induced Atelectasis in Patients Undergoing General Anesthesia Accessed by Pulmonary Ultrasound：Study Protocol for a Randomized, Double-blinded Controlled Trial
Brief Title: Effects of Small-dose S-ketamine on Anesthesia-induced Atelectasis in Anesthetized Patients Accessed by Pulmonary Ultrasound
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20210106
Record Dates: First submitted 2021-02-02; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Atelectasis
Keywords: atelectasis; S-ketamine; ultrasound; RCT; protocol
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-ketamine group (Experimental)
  Interventions: Drug: S-ketamine
- saline group (Placebo Comparator)
  Interventions: Drug: normal saline group

INTERVENTIONS:
Drug: S-ketamine — Patients will receive the label-covered trial agent covered by the label after premedication 5 min before induction. Agent preparation method of S-ketamine group (Group S): Draw the dosage of S-ketamine 0.25mg ·kg -1 and dilute it with normal saline to 5ml in opaque 5-ml syringes.
  Arms: S-ketamine group
Drug: normal saline group — Patients will receive the label-covered trial agent covered by the label after premedication 5 min before induction. Normal saline group (Group N): 5ml of normal saline, labeled as "study agents".
  Arms: saline group

SUMMARY:
Background: Atelectasis occurs in the majority of patients with general anesthesia, which can lead to postoperative pulmonary complications (PPCs) and affect the postoperative outcome. However, there is still no exact method to prevent it though agents. S-ketamine may prevent atelectasis due to its airway smooth muscle relaxation and anti-inflammatory effects. Lung ultrasound is a portable and reliable bedside imaging technology for diagnosing anesthesia-induced atelectasis. Here, we intend to assess whether small-dose of S-ketamine can reduce the incidence of atelectasis after intubation under general anesthesia using lung ultrasound, in order to prevent the early formation of perioperative atelectasis and perioperative pulmonary complications.

Methods: The trial is a single institution, prospective, randomized controlled, parallel grouping, double-blind study. From October 2021 to March 2022, 100 patients (18-60 years old) scheduled for elective surgery will be recruited from Beijing Tiantan Hospital, Capital Medical University, and randomly assigned to the S-ketamine group (Group S) and the normal saline group (Group N) at a ratio of 1:1. The label-masked agents will be given 5 minutes before induction and all patients will undergo a standardized general anesthesia protocol. Related data will be collected at three time point: after radial artery puncture (T1), 15 minutes after tracheal intubation (T2) and before extubation (T3). The primary outcome will be the total LUS scores at T2. Secondary outcomes include LUS scores in 6 chest regions at T2; total LUS scores at T3; arterial blood-gas analysis results (PaCO2, PaO2) and PaO2/FiO2 at T2 and T3, plateau pressure(Pplat) and dynamic lung compliance (Cdyn) at T2 and T3; the incidence of postoperative complications associated with S-ketamine and postoperative pulmonary complications (PPCs) 2 and 24 hours after surgery；.

Discussion: This trial aims to explore whether a simple and feasible application of S-ketamine before the induction of general anesthesia can prevent atelectasis. The results of this study may provide new ideas and direct clinical evidence for the prevention and treatment of perioperative pulmonary complications during anesthesia.

Key words: atelectasis, S-ketamine, ultrasound, RCT, protocol

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 - 60 years;
2. American Society of Anesthesiologists (ASA) physical status of I - II;
3. Patients scheduled for urinary, obstetrics and gynecology surgery in supine position or lithotomy position under general anesthesia, and the expected operation time is more than 1 hour;
4. Patients and their authorized surrogates have signed the informed consent form.

Exclusion Criteria:

1. Patients who have difficulty in applying pulmonary ultrasound, such as chest fractures, surgical history, etc;
2. Patients who have a history of upper respiratory tract infection one month before surgery, or a history of smoking more than 6 packs/year;
3. Preoperative chest X-ray or CT abnormalities, including atelectasis, pneumothorax, pleural effusion or pneumonia;
4. BMI>30kg/㎡;
5. Expected difficulty in intubation or mask ventilation;
6. Patients with significant increase in intraocular pressure and intracranial pressure before surgery;
7. Patients allergic to S-ketamine, propofol and opioids.
8. Patients with a positive history of psychiatric disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
total lung sonography scores(LUS) scores at T2 | T2：at the time of tracheal intubation
  Using SonoSite M-Turbo with a 5-12 MHz linear transducer,patients will be scanned and scored in the supine position following the lung ultrasound method described by Sun L and colleagues. Briefly, six regions will be scanned on in each hemithorax. Scans 1 and 2 will be performed at the midline of the clavicle, scans 3 and 4 will be performed in the axilla midline. The intercostal scans (Scans 5-6) will be performed in the fifth and sixth intercostal spaces of the posterior axillary line. Place a linear probe parallel to the ribs and scan the intercostal space of each region using a two-dimensional view sequentially from right to left, cranial to caudal, and anterior to posterior within 2 minutes.Each region will be categorised and assigned into four scores(0-3) based on B-lines.Add the scores in all twelve regions to get total lung sonography scores(LUS). Finally get a score between 0 (no atelectasis) and 36 (complete atelectasis).

SECONDARY OUTCOMES:
LUS scores in 6 chest regions(scans 1-6) at T2 | T2：at the time of tracheal intubation
  Using SonoSite M-Turbo with a 5-12 MHz linear transducer,patients will be scanned and scored in the supine position following the lung ultrasound method described by Sun L and colleagues. Briefly, six regions will be scanned on in each hemithorax. Scans 1 and 2 will be performed at the midline of the clavicle, scans 3 and 4 will be performed in the axilla midline. The intercostal scans (Scans 5-6) will be performed in the fifth and sixth intercostal spaces of the posterior axillary line. Place a linear probe parallel to the ribs and scan the intercostal space of each region using a two-dimensional view sequentially from right to left, cranial to caudal, and anterior to posterior within 2 minutes.Each region will be categorised and assigned into four scores(0-3) based on B-lines. Finally get six sets of data betweem 0(no atelectasis) and 6 (complete atelectasis).
total LUS scores at T3 | T3：5min before extubation
  Using SonoSite M-Turbo with a 5-12 MHz linear transducer,patients will be scanned and scored in the supine position following the lung ultrasound method described by Sun L and colleagues. Briefly, six regions will be scanned on in each hemithorax. Scans 1 and 2 will be performed at the midline of the clavicle, scans 3 and 4 will be performed in the axilla midline. The intercostal scans (Scans 5-6) will be performed in the fifth and sixth intercostal spaces of the posterior axillary line. Place a linear probe parallel to the ribs and scan the intercostal space of each region using a two-dimensional view sequentially from right to left, cranial to caudal, and anterior to posterior within 2 minutes.Each region will be categorised and assigned into four scores(0-3) based on B-lines. Finally get a score between 0 (no atelectasis) and 36 (complete atelectasis).
arterial blood-gas analysis results (PaCO2, PaO2) and PaO2/FiO2 at T2 and T3 | after tracheal intubation (T2) and 5min before extubation (T3)
  arterial blood samples will be obtained through radial artery puncture and blood-gas measurements will be performed immediately using a standard technique (ABL800) to get arterial blood-gas analysis results (PaCO2, PaO2) and PaO2/FiO2 at T2 and T3
plateau pressure and dynamic lung compliance (Cdyn) at T2 and T3 | after tracheal intubation (T2) and 5min before extubation (T3)
  [Cdyn = tidal volume/(PIP-PEEP)]
the incidence of postoperative complications associated with S-ketamine 2 and 24 hours after surgery | 2 and 24 hours after surgery
  visual impairment, dizziness, pathological irritability, nightmares and hallucinations
the incidence of postoperative pulmonary complications (PPCs) | 2 and 24 hours after surgery
  the clinical outcome defifinitions of PPCs will adopt European joint taskforce guidelines published in 2015 which include respiratory infection; respiratory failure; atelectasis; pleural effusion; pneumothorax; bronchospasm, aspiration pneumonia; pulmonary edema; ARDS; tracheobronchitis; pulmonary oedema; exacerbation of pre-existing lung disease; pulmonary embolism

REFERENCES:
- [Derived] Zhang D, Liang Y, Bao D, Xiong W, Li L, Wang Y, Liu B, Jin X. Effects of small-dose S-ketamine on anesthesia-induced atelectasis in patients undergoing general anesthesia accessed by lung ultrasound: study protocol for a randomized, double-blinded controlled trial. Trials. 2024 Jan 18;25(1):64. doi: 10.1186/s13063-023-07779-y. PMID 38238838